CLINICAL TRIAL: NCT06136559
Title: A Phase 3, Randomized Study to Compare Nemtabrutinib Versus Comparator (Investigator's Choice of Ibrutinib or Acalabrutinib) in Participants With Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (BELLWAVE-011)
Brief Title: A Study of Nemtabrutinib (MK-1026) Versus Comparator (Investigator's Choice of Ibrutinib or Acalabrutinib) in First Line (1L) Chronic Lymphocytic Leukemia (CLL)/ Small Lymphocytic Lymphoma (SLL) (MK-1026-011/BELLWAVE-011)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026-011; 2022-501697-19-00 (Registry Identifier: EU CT); U1111-1281-7895 (Registry Identifier: UTN); MK-1026-011 (Other: MSD); BELLWAVE-011 (Other: MSD); jRCT2031230697 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ARQ531; ibrutinib; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemtabrutinib (Experimental): Participants will receive nemtabrutinib at specified dose until disease progression, unacceptable toxicity or until discontinuation criteria are met.
  Interventions: Drug: Nemtabrutinib
- Ibrutinib/Acalabrutinib (Active Comparator): Participants will receive investigator's choice of ibrutinib or acalabrutinib at specified dose until disease progression, unacceptable toxicity or until discontinuation criteria are met.
  Interventions: Drug: Ibrutinib; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Administered orally
  Other Names: MK-1026; ARQ 531
  Arms: Nemtabrutinib
Drug: Ibrutinib — Administered orally
  Arms: Ibrutinib/Acalabrutinib
Drug: Acalabrutinib — Administered orally
  Arms: Ibrutinib/Acalabrutinib

SUMMARY:
The goal of this study is to evaluate nemtabrutinib compared with investigator's choice of ibrutinib or acalabrutinib in participants with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) who have not received any prior therapy. The primary hypotheses are that (1) nemtabrutinib is non-inferior to ibrutinib or acalabrutinib with respect to objective response rate (ORR) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria 2018 by blinded independent central review (BICR) and (2) nemtabrutinib is superior to ibrutinib or acalabrutinib with respect to progression free survival (PFS) per iwCLL Criteria 2018 by BICR.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Confirmed diagnosis of CLL/SLL and active disease clearly documented to have a need to initiate therapy.
* Has at least 1 marker of disease burden.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 within 7 days before randomization.
* Has the ability to swallow and retain oral medication.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV deoxyribonucleic acid (DNA) viral load before randomization.
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV ribonucleic acid (RNA) viral load is undetectable at screening.
* Participants with human immunodeficiency virus (HIV) who meet ALL eligibility criteria.

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has an active hepatitis B virus/ hepatitis C virus (HBV/HCV) infection.
* Has gastrointestinal (GI) dysfunction that may affect drug absorption.
* Has diagnosis of Richter Transformation or active central nervous system (CNS) involvement by CLL/SLL.
* Has had acquired immune deficiency syndrome (AIDS)-defining opportunistic infection in the past 12 months before screening.
* Has clinically significant cardiovascular disease.
* Has hypersensitivity to nemtabrutinib or contraindication to ibrutinib or acalabrutinib, or any of the excipients.
* Has history of severe bleeding disorder.
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Has received any systemic anticancer therapy for CLL/SLL.
* Is currently being treated with p-glycoprotein (P-gp) substrates with a narrow therapeutic index, cytochrome P450 3A (CYP3A) strong or moderate inducers or CYP3A strong inhibitors.
* Received prior radiotherapy within 2 weeks of start of study intervention, or radiation-related toxicities, requiring corticosteroids.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks before study intervention administration.
* Has active infection requiring systemic therapy, including intravenous (IV) antibiotics during screening.
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2032-09-07 (Estimated); Study Completion 2032-09-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per Chronic Lymphocytic Leukemia (iwCLL) Criteria 2018 as assessed by Blinded Independent Central Review (BICR) | Up to ~33 months
  ORR is defined as the percentage of participants with complete response (CR), complete response with an incomplete recovery of the participant's bone marrow (CRi), nodular partial response (nPR), or partial response (PR), per iwCLL Criteria 2018 as assessed by BICR.
Progression-Free Survival (PFS) per iwCLL Criteria 2018 as assessed by BICR | Up to ~104 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PD is evaluated per iwCLL Criteria 2018 as assessed by BICR.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~104 months
  OS is defined as the time from randomization to death due to any cause.
Duration of Response (DOR) per iwCLL Criteria 2018 as assessed by BICR | Up to ~104 months
  For participants who demonstrate a complete response (CR), complete response with an incomplete recovery of the participant's bone marrow (CRi), nodular partial response (nPR), or partial response (PR) per iwCLL Criteria 2018 as assessed by BICR, DOR is defined as the time from the first documented evidence of CR, CRi, nPR, or PR that led to response until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to ~104 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to ~104 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (194):
- United States (39):
  - USA Mitchell Cancer Institute ( Site 0014), Mobile, Alabama
  - Banner MD Anderson Cancer Center - University Medical Center Phoenix ( Site 0051), Phoenix, Arizona
  - Arizona Oncology Associates - NAHOA ( Site 8007), Prescott, Arizona
  - Alta Bates Summit Medical Center ( Site 0004), Berkeley, California
  - Moores Cancer Center ( Site 0003), La Jolla, California
  - Saint Joseph Hospital ( Site 0026), Denver, Colorado
  - Lutheran Medical Center ( Site 0027), Golden, Colorado
  - Intermountain Health St. Mary's Regional Hospital ( Site 0025), Grand Junction, Colorado
  - Eastern CT Hematology & Oncology Associates ( Site 0033), Norwich, Connecticut
  - Clermont Oncology Center ( Site 0046), Clermont, Florida
  - Florida Cancer Specialists - South ( Site 7001), Fort Myers, Florida
  - Florida Cancer Specialists - East ( Site 7002), West Palm Beach, Florida
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0002), Fort Wayne, Indiana
  - University of Iowa Health Care. ( Site 0017), Waukee, Iowa
  - University of Iowa Health Care. ( Site 0057), Waukee, Iowa
  - Saint Elizabeth Healthcare ( Site 0041), Edgewood, Kentucky
  - Corewell Health-Lemmon Holton Cancer Pavilion ( Site 0011), Grand Rapids, Michigan
  - Regions Hospital ( Site 0042), Saint Louis Park, Minnesota
  - MidAmerica Cancer Care, LLC ( Site 0043), Kansas City, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana ( Site 0052), Billings, Montana
  - Summit Medical Group Cancer Center ( Site 0007), Florham Park, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0016), Hackensack, New Jersey
  - Roswell Park Cancer Institute ( Site 0023), Buffalo, New York
  - Oncology Specialists of Charlotte ( Site 0054), Charlotte, North Carolina
  - Southeastern Medical Oncology Center ( Site 0049), Goldsboro, North Carolina
  - Consultants in Medical Oncology and Hematology (CMOH) ( Site 8002), Broomall, Pennsylvania
  - Cancer Care Associates Of York ( Site 0005), York, Pennsylvania
  - Tennessee Oncology-Chattanooga ( Site 0045), Chattanooga, Tennessee
  - Tennessee Oncology, PLLC - Elliston Place Plaza Medical Oncology & Hematology ( Site 0031), Nashville, Tennessee
  - Texas Oncology - Central/South Texas ( Site 8008), Austin, Texas
  - The Center for Cancer and Blood Disorders ( Site 0032), Fort Worth, Texas
  - Texas Oncology - San Antonio ( Site 8006), San Antonio, Texas
  - Texas Oncology - Northeast Texas ( Site 8012), Tyler, Texas
  - University of Virginia Cancer Center ( Site 0040), Charlottesville, Virginia
  - Inova Schar Cancer Institute ( Site 0015), Fairfax, Virginia
  - Virginia Commonwealth University (VCU) Medical Center ( Site 0030), Richmond, Virginia
  - Medical Oncology Associates, PS (dba Summit Cancer Centers) ( Site 0010), Spokane, Washington
  - SSM Health Dean Medical Group - South Madison Campus Health Research/Circuit Clinical ( Site 0048), Madison, Wisconsin
  - University Hospital and UW Health Clinics ( Site 0006), Madison, Wisconsin
- Royal North Shore Hospital ( Site 2806), St Leonards, New South Wales, Australia
- Belgium (2):
  - AZ Sint-Maarten, Campus Leopoldstraat 2 ( Site 0205), Mechelen, Antwerpen
  - UZ Leuven-Hematology ( Site 0200), Leuven, Vlaams-Brabant
- Brazil (3):
  - Hospital 9 De Julho ( Site 2206), São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 2201), Rio de Janeiro
  - Hospital Paulistano-Americas Oncologia ( Site 2202), São Paulo
- Canada (6):
  - BC Cancer Kelowna ( Site 0112), Kelowna, British Columbia
  - BC Cancer Victoria ( Site 0109), Victoria, British Columbia
  - William Osler Health System ( Site 0103), Brampton, Ontario
  - The Ottawa Hospital - General Campus ( Site 0102), Ottawa, Ontario
  - McGill University Health Centre ( Site 0106), Montreal, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski ( Site 0100), Rimouski, Quebec
- Chile (3):
  - FALP-UIDO ( Site 2300), Santiago, Region M. de Santiago
  - Clínica Alemana de Santiago-Unidad de Investigaciones ( Site 2306), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 2310), Santiago, Region M. de Santiago
- China (30):
  - Anhui Provincial Cancer Hospital ( Site 2001), Hefei, Anhui
  - Peking University First Hospital ( Site 2022), Beijing, Beijing Municipality
  - Peking University Third Hospital-Hematology ( Site 2011), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 2041), Chongqing, Chongqing Municipality
  - Southern Medical University Nanfang Hospital-Department of Hematopathology ( Site 2006), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 2028), Guangzhou, Guangdong
  - Liuzhou People's Hospital ( Site 2029), Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 2004), Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University ( Site 2024), Guiyang, Guizhou
  - Hainan General Hospital ( Site 2018), Haikou, Hainan
  - Wuhan Union Hospital ( Site 2015), Wuhan, Hebei
  - Henan Cancer Hospital-hematology department ( Site 2025), Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of HUST ( Site 2016), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 2020), Changsha, Hunan
  - The Second Xiangya Hospital of Central South University ( Site 2010), Changsha, Hunan
  - Jiangsu Province Hospital ( Site 2000), Nanjing, Jiangsu
  - The First Affliated Hospital of Suzhou University ( Site 2027), Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 2013), Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 2023), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 2009), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 2030), Changchun, Jilin
  - Shaanxi provincial people's hospital ( Site 2012), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 2003), Jinan, Shandong
  - Shanxi Cancer Hospital ( Site 2033), Taiyuan, Shanxi
  - West China Hospital, Sichuan University-Head and Neck Oncology ( Site 2026), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital-lymphoma ( Site 2019), Tianjin, Tianjin Municipality
  - Institute of hematology&blood disease hospital-Lymphoma ( Site 2005), Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 2014), Ürümqi, Xinjiang
  - The first Affiliated Hospital, Zhejiang University School of Medicine-Hematology ( Site 2002), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2017), Hangzhou, Zhejiang
- Colombia (3):
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 2405), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 2401), Montería, Departamento de Córdoba
  - Fundacion Valle del Lili- CIC-Oncology CIC ( Site 2402), Cali, Valle del Cauca Department
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove-IV. interni hematologicka klinika ( Site 0301), Hradec Králové
  - Fakultni nemocnice Olomouc ( Site 0303), Olomouc
  - Vseobecna fakultni nemocnice v Praze-I. Interní klinika - klinika hematologie ( Site 0302), Prague
- Denmark (3):
  - Aalborg Universitetshospital, Syd ( Site 0403), Aalborg, North Denmark
  - Roskilde Sygehus-Department of Hematology ( Site 0402), Roskilde, Region Sjælland
  - Odense Universitetshospital-Department of Hematology ( Site 0401), Odense C, Region Syddanmark
- Germany (6):
  - Universitaetsklinikum Ulm. ( Site 0601), Ulm, Baden-Wurttemberg
  - VK&K Studien GbR ( Site 0607), Landshut, Bavaria
  - Kliniken Maria Hilf ( Site 0603), Mönchengladbach, North Rhine-Westphalia
  - InVO Institut für Versorgungsforschung in der Onkologie ( Site 0606), Koblenz, Rhineland-Palatinate
  - Universitätsklinikum Halle ( Site 0604), Halle, Saxony-Anhalt
  - Onkologische Schwerpunktpraxis Kurfuerstendamm ( Site 0600), Berlin
- Greece (4):
  - Evangelismos General Hospital of Athens ( Site 0700), Athens, Attica
  - General Hospital of Athens "Laiko" ( Site 0704), Athens, Attica
  - University Hospital of Alexandroupolis ( Site 0701), Alexandroupoli, East Macedonia and Thrace
  - University Hospital of Ioannina ( Site 0702), Ioannina
- Queen Mary Hospital ( Site 3300), Hong Kong, Hong Kong
- Israel (7):
  - Rambam Health Care Campus-Hematology and Bone Marrow Transplantation ( Site 1503), Haifa
  - Bnai Zion Medical Center ( Site 1505), Haifa
  - Hadassah Medical Center-Hemato-Oncology ( Site 1500), Jerusalem
  - Galilee Medical Center ( Site 1507), Nahariya
  - Rabin Medical Center ( Site 1504), Petah Tikva
  - Sheba Medical Center-Hemato Oncology ( Site 1501), Ramat Gan
  - Yitzhak Shamir Medical Center. ( Site 1506), Ẕerifin
- Japan (14):
  - Nagoya University Hospital ( Site 1907), Nagoya, Aichi-ken
  - Gunma University Hospital ( Site 1903), Maebashi, Gunma
  - Hokkaido University Hospital ( Site 1900), Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital ( Site 1910), Kobe, Hyōgo
  - Tohoku University Hospital ( Site 1901), Sendai, Miyagi
  - Kindai University Hospital ( Site 1909), Sakai, Osaka
  - Shimane University Hospital ( Site 1911), Izumo, Shimane
  - Cancer Institute Hospital of JFCR ( Site 1906), Koto, Tokyo
  - Chiba Cancer Center ( Site 1905), Chiba
  - Kyushu University Hospital ( Site 1914), Fukuoka
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital ( Site 1913), Hiroshima
  - Okayama University Hospital ( Site 1912), Okayama
  - Japanese Red Cross Osaka Hospital ( Site 1908), Osaka
  - Yamagata University Hospital ( Site 1902), Yamagata
- Malaysia (3):
  - University Malaya Medical Centre ( Site 1604), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 1602), George Town, Pulau Pinang
  - Queen Elizabeth Hospital ( Site 1603), Kota Kinabalu, Sabah
- Mexico (3):
  - Centro de Infusion Superare ( Site 2602), Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V: ( Site 2608), Mexico City, Mexico City
  - Grupo Médico ASSET ( Site 2611), Mexico City
- New Zealand (3):
  - Waikato Hospital-Haematology ( Site 3202), Hamilton, Waikato Region
  - North Shore Hospital-Department of Haematology ( Site 3200), Auckland
  - Aotearoa Clinical Trials ( Site 3201), Auckland
- Norway (3):
  - Akershus Universitetssykehus ( Site 0902), Lørenskog, Akershus
  - Sykehuset i Vestfold ( Site 0903), Tønsberg, Vestfold
  - Oslo Universitetssykehus Rikshospitalet-Avdeling for blodsykdommer ( Site 0901), Oslo
- Peru (2):
  - Centro Medico Monte Carmelo-Oncology ( Site 2706), Arequipa, Ariqipa
  - Clínica Anglo Americana ( Site 2701), Lima
- Poland (8):
  - Pratia MCM Krakow ( Site 1007), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 1 w Lublinie-Oddział Hematoonkologii-Transplantacji Szpiku i Chem ( Site 1006), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Kilinka Onkologii I Hematologii ( Site 1004), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 1011), Gdansk, Pomeranian Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. J. Korczaka w Słupsku-Oddział Hematologii i Transplantacji ( Site 1013), Słupsk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 1000), Gliwice, Silesian Voivodeship
  - Pratia Onkologia Katowice ( Site 1009), Katowice, Silesian Voivodeship
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej MSWiA w Olsztynie-Oddzial Kliniczny Hematologii ( Site 1005), Olsztyn, Warmian-Masurian Voivodeship
- Portugal (6):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil ( Site 3103), Lisbon, Lisbon District
  - Champalimaud Foundation ( Site 3102), Lisbon, Lisbon District
  - Unidade Local de Saude Gaia/Espinho - Hospital Eduardo Santos Silva ( Site 3107), Vila Nova de Gaia, Porto District
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 3104), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 3106), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 3100), Porto
- South Africa (5):
  - Wits Clinical Research ( Site 1102), Johannesburg, Gauteng
  - Netcare Pretoria East Hospital-Alberts Cellular Therapy ( Site 1101), Pretoria, Gauteng
  - Groote Schuur Hospital-Clinical Haematology ( Site 1100), Cape Town, Western Cape
  - Haemalife ( Site 1105), Kuilsriver, Western Cape
  - Constantiaberg Haematology ( Site 1106), Plumstead, Western Cape
- Spain (7):
  - Institut Català d'Oncologia - L'Hospitalet-Haematology Department ( Site 1207), L'Hospitalet Del Llobregat, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 1202), Barcelona, Catalonia
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 1209), Pozuelo de Alarcón, Madrid
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA ( Site 1208), Majadahonda, Madrid, Comunidad de
  - hospital universitario de canarias ( Site 1205), San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1206), Barcelona
  - Hospital Universitario de Salamanca - Complejo Asistencial U-Servicio de Hematologia ( Site 1201), Salamanca
- Karolinska Universitetssjukhuset Solna ( Site 1302), Stockholm, Stockholm County, Sweden
- Taiwan (4):
  - Chang Gung Memorial Hospital at Kaohsiung-Division of Hematology and Oncology ( Site 1702), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 1700), Tainan
  - National Taiwan University Hospital ( Site 1701), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 1703), Taoyuan District
- Thailand (5):
  - Chulalongkorn University ( Site 1802), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Division of Hematology, Department of Medicine ( Site 1801), Bangkok, Bangkok
  - Naresuan University Hospital ( Site 1804), Muang, Changwat Phitsanulok
  - Songklanagarind hospital ( Site 1803), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 1800), Muang, Chiang Mai
- Turkey (Türkiye) (9):
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 1401), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1407), Ankara
  - Antalya Egitim ve Arastırma Hastanesi ( Site 1409), Antalya
  - Trakya University Medical Faculty Hospital-Hematology ( Site 1403), Edirne
  - Mega Medipol ( Site 1412), Istanbul
  - Sisli Florence Nightingale Hastanesi ( Site 1411), Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi ( Site 1408), Istanbul
  - Ege Universitesi Hastanesi ( Site 1404), Izmir
  - Ondokuz Mays Üniversitesi ( Site 1410), Samsun
- United Kingdom (10):
  - Southmead Hospital ( Site 3010), Bristol, Bristol, City of
  - Royal Lancaster Infirmary ( Site 3012), Lancaster, Lancashire
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 3006), London, London, City of
  - The Churchill Hospital ( Site 3007), Oxford, Oxfordshire
  - GenesisCare - Bristol ( Site 3011), Bristol, South Gloucestershire
  - GenesisCare - Cambridge ( Site 3001), Newmarket, Suffolk
  - GenesisCare - Windsor ( Site 3002), Windsor, Windsor And Maidenhead
  - Barnet Hospital ( Site 3005), Barnet
  - St James's University Hospital ( Site 3004), Leeds
  - City Hospital, Nottingham University Hospitals NHS Trust ( Site 3003), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26310&tenant=MT_MSD_9011